CLINICAL TRIAL: NCT03061331
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy of Lumacaftor/Ivacaftor Combination Therapy in Subjects With Cystic Fibrosis Who Have an A455E-CFTR Mutation
Brief Title: Lumacaftor/Ivacaftor Combination Therapy in Subjects With CF Who Have an A455E CFTR Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15-809-111; 2016-001585-29 (EudraCT Number)
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence 1 (Experimental): LUM/IVA in Treatment Period 1; washout; placebo in Treatment Period 2
  Interventions: Drug: LUM/IVA; Drug: Placebo
- Treatment Sequence 2 (Experimental): Placebo in Treatment Period 1; washout; LUM/IVA in Treatment Period 2
  Interventions: Drug: LUM/IVA; Drug: Placebo

INTERVENTIONS:
Drug: LUM/IVA — LUM 400 mg/IVA 250 mg every 12 hours (q12h)
  Other Names: lumacaftor/ivacaftor
Drug: Placebo — No Active Drug

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter, crossover study that will evaluate the efficacy of LUM/IVA in subjects with CF 12 years of age and older who have at least one A455E mutation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF
* All subjects must have an A455E mutation on at least 1 CFTR allele; no more than 10 subjects may have an F508del mutation on 1 CFTR allele.
* Forced expiratory volume in one second (FEV1) ≥30% of predicted and ≤90% of predicted at the Screening Visit, based on the Global Lung Function Initiative (GLI)-2012 multi ethnic all-age reference equations.
* Stable CF disease as judged by the investigator.
* Willing to remain on a stable medication regimen for CF from 4 weeks before Day 1 through the Follow up Visit.

Exclusion Criteria:

* History of any comorbidity reviewed at the Screening Visit that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* A G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, S549R, or R117H mutation on at least one CFTR allele.
* Pregnant or breastfeeding.
* Any abnormal laboratory values at the Screening Visit.
* History of cataract/lens opacity, or evidence of cataract/lens opacity determined to be clinically significant by the ophthalmologist or optometrist during the ophthalmologic examination at the Screening Visit.
* Use of strong inhibitors or strong inducers of CYP3A, including consumption of certain herbal medications and certain fruit and fruit juices, within 14 days before Day 1
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - HagaZiekenhuis, The Hague

REFERENCES:
- [Derived] Berkers G, van der Meer R, Heijerman H, Beekman JM, Boj SF, Vries RGJ, van Mourik P, Doyle JR, Audhya P, Yuan ZJ, Kinnman N, van der Ent CK. Lumacaftor/ivacaftor in people with cystic fibrosis with an A455E-CFTR mutation. J Cyst Fibros. 2021 Sep;20(5):761-767. doi: 10.1016/j.jcf.2020.11.007. Epub 2020 Nov 26. PMID 33249003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 subjects were enrolled in this cross-over study.
Groups:
- Sequence 1: First LUM/IVA, Then Placebo: Participants received Lumacaftor (LUM) 400 milligram (mg)/Ivacaftor (IVA) 250 mg fixed dose combination tablet orally every 12 hours (q12h) for 8 weeks in treatment period 1 followed by placebo matched to LUM/IVA tablet orally q12h for 8 weeks in treatment period 2. Two treatment periods were separated by 8-week washout period.
- Sequence 2: First Placebo, Then LUM/IVA: Participants received placebo matched to LUM/IVA tablet orally q12h for 8 weeks in treatment period 1 followed by LUM 400 mg/IVA 250 mg fixed dose combination tablet orally q12h for 8 weeks in treatment period 2. Two treatment periods were separated by 8-week washout period.
Period: Treatment Period 1 (8 Weeks)
Arm/Group | Sequence 1: First LUM/IVA, Then Placebo | Sequence 2: First Placebo, Then LUM/IVA
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period (8 Weeks)
Arm/Group | Sequence 1: First LUM/IVA, Then Placebo | Sequence 2: First Placebo, Then LUM/IVA
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Treatment Period 2 (8 Weeks)
Arm/Group | Sequence 1: First LUM/IVA, Then Placebo | Sequence 2: First Placebo, Then LUM/IVA
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: First LUM/IVA, Then Placebo: Participants received LUM 400 mg/IVA 250 mg fixed dose combination tablet orally q12h for 8 weeks in treatment period 1 followed by placebo matched to LUM/IVA tablet orally q12h for 8 weeks in treatment period 2. Two treatment periods were separated by 8-week washout period.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: First LUM/IVA, Then Placebo | Sequence 2: First Placebo, Then LUM/IVA | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (15.1) | 34.7 (11.8) | 38.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Through Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Study Baseline, Through Week 8
Population: Full Analysis set included as all randomized participants who had at least 1 A455E mutation and received at least 1 dose of study drug. Here "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FEV1
Groups:
- Placebo: Placebo matched to LUM/IVA q12h for 8 weeks in Treatment Period 1 or 2
- LUM/IVA: LUM 400 mg/IVA 250 mg fixed dose combination q12h for 8 weeks in Treatment Period 1 or 2.
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 18 | 18
Percentage of predicted FEV1 | 2.6 [0.2 to 4.9] | 2.7 [0.3 to 5.0]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.9277, Mixed Model Repeated Measure (MMRM); Least Squares Mean Difference = 0.1, 95% CI 2-sided [-2.5 to 2.7]

ADVERSE EVENTS:
Time Frame: Up to Week 28
Arm/Group | Placebo | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 13/18 | 15/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | LUM/IVA (N=19)
Hypertension (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 2 | 3
Exercise tolerance decreased (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 8
Flatulence (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 2
Herpes zoster (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03061331/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03061331/SAP_001.pdf